CLINICAL TRIAL: NCT01078402
Title: Evaluation of Clinical Outcome, Treatment Compliance and Tolerability of humIRA (Adalimumab) in Patients With Active Rheumatoid Arthritis, Psoriatic Arthritis and Ankylosing Spondylitis in EASTern European Countries; EviraEAST - a Multi-country, Multi-Center Post Marketing Observational Study in Routine Clinical Use
Brief Title: EValuation of HumIRA® in Patients With Active Rheumatoid Arthritis, Psoriatic Arthritis and Ankylosing Spondylitis in EASTern European Countries
Acronym: EviraEAST
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P10-919
Record Dates: First submitted 2010-02-27; First posted 2010-03-02 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Ankylosing Spondylitis (AS); Psoriatic Arthritis (PsA; Rheumatoid Arthritis (RA
Keywords: Treatment compliance and tolerability of Humira in patients; Eastern European countries; Rheumatoid Arthritis; Psoriatic Arthritis; Adalimumab; Ankylosing Spondylitis; Evaluation of clinical outcome
MeSH Terms: conditions — Spondylitis, Ankylosing; Arthritis, Psoriatic; Salivary Gland Adenoma, Pleomorphic; Arthritis, Rheumatoid; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single patients group: RA, PsA and AS: Single patients group with: Active Rheumatoid Arthritis (RA), Psoriatic Arthritis (PsA) and Ankylosing Spondylitis (AS)

SUMMARY:
This is a non-interventional, post-marketing, observational study (PMOS) in which Humira (adalimumab) is prescribed in the usual manner in accordance with the terms of the local marketing authorization with regards to dose, population and indication. No data currently exists to characterize patient populations being prescribed Humira in Eastern Europe. Further, it is important to establish the clinical outcome and tolerability of Humira in Eastern European patients, as well as their compliance with Humira treatment, in particular the acceptability of self-injection, which may influence all of the above in routine clinical practice.

DETAILED DESCRIPTION:
This PMOS will be conducted in a prospective, single-arm, multicountry, multicenter format. The assignment of the patient to Humira is not decided in advance by this protocol but falls within the current practice. The prescription of Humira is clearly separated from the decision to include the patient in this study. No additional procedures (other than standard of care) shall be applied to the patients. As this study is observational in nature, its follow-up is not interventional and is left to the judgment of each physician within the 14-17 months period (including tuberculosis (TB) screening and prophylaxis, if indicated), which defines the survey for each patient. The TB screening period per patient will be 1-4 weeks and, if applicable, the TB prophylactic treatment period before Humira administration will be 1 month in accordance with local guidelines. For indicative purposes, follow-up of patients should entail approximately 7 patient visits during this period. These visits will take place at average intervals of 3 months, apart from the first visit following TB screening. The first visit following introduction of Humira and final visits are required because of intercurrent events. If treatment with Humira is discontinued, the standard practice is to review the patient after a period of 70 days or 5 half-lives following the intake of the last dose of physician-prescribed treatment. If the physician decides to permanently discontinue Humira before the end of the planned observational period of 13 months, the reason for discontinuation and the new treatment regimen prescribed, if applicable, will be documented. The next routine follow-up visit will be the termination visit for this patient in the PMOS.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients with active RA, PsA or AS for whom Humira therapy is indicated according to the local product label and who meet the following criteria:

* Are newly prescribed Humira therapy (no prior history of treatment with Humira), including patients with infliximab or etanercept treatment history OR
* Completed Abbott sponsored interventional clinical trials and are continuing treatment with commercial Humira thereafter.

Exclusion Criteria:

* Patients who are being treated or will be treated with drugs at risk of interactions with Humira (see Humira Summary of Product Characteristics)
* Patients currently participating in another clinical trial
* Patients with diagnosis of active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of adult patients in Eastern European countries with rheumatoid arthritis (RA), psoriatic arthritis (PsA) or ankylosing spondylitis (AS) who can be administered Humira as per locally approved label.
Sampling Method: Non-Probability Sample
Enrollment: 809 (Actual)
Dates: Start 2009-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maja Hojnik, Study Director — AbbVie
Locations (163):
- Croatia (6):
  - Site Reference ID/Investigator# 43283, Opatija
  - Site Reference ID/Investigator# 43282, Osijek
  - Site Reference ID/Investigator# 43286, Rijeka
  - Site Reference ID/Investigator# 43284, Split
  - Site Reference ID/Investigator# 22405, Zagreb
  - Site Reference ID/Investigator# 43285, Zagreb
- Hungary (71):
  - Site Reference ID/Investigator# 32641, Budapest
  - Site Reference ID/Investigator# 32642, Budapest
  - Site Reference ID/Investigator# 32676, Budapest
  - Site Reference ID/Investigator# 32677, Budapest
  - Site Reference ID/Investigator# 32679, Budapest
  - Site Reference ID/Investigator# 32680, Budapest
  - Site Reference ID/Investigator# 32681, Budapest
  - Site Reference ID/Investigator# 32682, Budapest
  - Site Reference ID/Investigator# 32685, Budapest
  - Site Reference ID/Investigator# 32686, Budapest
  - Site Reference ID/Investigator# 32687, Budapest
  - Site Reference ID/Investigator# 32688, Budapest
  - Site Reference ID/Investigator# 32689, Budapest
  - Site Reference ID/Investigator# 32691, Budapest
  - Site Reference ID/Investigator# 32692, Budapest
  - Site Reference ID/Investigator# 32693, Budapest
  - Site Reference ID/Investigator# 32633, Budapest
  - Site Reference ID/Investigator# 32634, Budapest
  - Site Reference ID/Investigator# 32635, Budapest
  - Site Reference ID/Investigator# 32636, Budapest
  - Site Reference ID/Investigator# 32638, Budapest
  - Site Reference ID/Investigator# 32639, Budapest
  - Site Reference ID/Investigator# 32640, Budapest
  - Site Reference ID/Investigator# 32694, Budapest
  - Site Reference ID/Investigator# 32695, Budapest
  - Site Reference ID/Investigator# 32612, Debrecen
  - Site Reference ID/Investigator# 32613, Debrecen
  - Site Reference ID/Investigator# 32614, Debrecen
  - Site Reference ID/Investigator# 32615, Debrecen
  - Site Reference ID/Investigator# 32616, Debrecen
  - Site Reference ID/Investigator# 32591, Debrecen
  - Site Reference ID/Investigator# 32592, Debrecen
  - Site Reference ID/Investigator# 32584, Esztergom
  - Site Reference ID/Investigator# 32585, Esztergom
  - Site Reference ID/Investigator# 32629, Győr
  - Site Reference ID/Investigator# 32630, Győr
  - Site Reference ID/Investigator# 32696, Gyula
  - Site Reference ID/Investigator# 32697, Gyula
  - Site Reference ID/Investigator# 32698, Gyula
  - Site Reference ID/Investigator# 32699, Gyula
  - Site Reference ID/Investigator# 32700, Gyula
  - Site Reference ID/Investigator# 32701, Gyula
  - Site Reference ID/Investigator# 32702, Gyula
  - Site Reference ID/Investigator# 32703, Gyula
  - Site Reference ID/Investigator# 32566, Hévíz
  - Site Reference ID/Investigator# 32580, Kecskemét
  - Site Reference ID/Investigator# 32581, Kecskemét
  - Site Reference ID/Investigator# 32582, Kistarcsa
  - Site Reference ID/Investigator# 32583, Kistarcsa
  - Site Reference ID/Investigator# 32624, Miskolc
  - Site Reference ID/Investigator# 32625, Miskolc
  - Site Reference ID/Investigator# 32626, Miskolc
  - Site Reference ID/Investigator# 32586, Nyíregyháza
  - Site Reference ID/Investigator# 32588, Nyíregyháza
  - Site Reference ID/Investigator# 32589, Nyíregyháza
  - Site Reference ID/Investigator# 32590, Nyíregyháza
  - Site Reference ID/Investigator# 32704, Pécs
  - Site Reference ID/Investigator# 32705, Pécs
  - Site Reference ID/Investigator# 32709, Pécs
  - Site Reference ID/Investigator# 32617, Szeged
  - Site Reference ID/Investigator# 32618, Szeged
  - Site Reference ID/Investigator# 32619, Szeged
  - Site Reference ID/Investigator# 32627, Székesfehérvár
  - Site Reference ID/Investigator# 32628, Székesfehérvár
  - Site Reference ID/Investigator# 32594, Szolnok
  - Site Reference ID/Investigator# 32595, Szolnok
  - Site Reference ID/Investigator# 32620, Szombathely
  - Site Reference ID/Investigator# 32622, Szombathely
  - Site Reference ID/Investigator# 32711, Veszprém
  - Site Reference ID/Investigator# 32712, Veszprém
  - Site Reference ID/Investigator# 32713, Veszprém
- Israel (6):
  - Site Reference ID/Investigator# 32079, Ashkelon
  - Site Reference ID/Investigator# 32082, Haifa
  - Site Reference ID/Investigator# 32080, Haifa
  - Site Reference ID/Investigator# 32081, Tel Litwinsky
  - Site Reference ID/Investigator# 65468, Tel Litwinsky
  - Site Reference ID/Investigator# 32078, Zrifin
- Poland (11):
  - Site Reference ID/Investigator# 32599, Bytom
  - Site Reference ID/Investigator# 43251, Krakow
  - Site Reference ID/Investigator# 32559, Krakow
  - Site Reference ID/Investigator# 32560, Krakow
  - Site Reference ID/Investigator# 43244, Krakow
  - Site Reference ID/Investigator# 43252, Krakow
  - Site Reference ID/Investigator# 43245, Poznan
  - Site Reference ID/Investigator# 43246, Poznan
  - Site Reference ID/Investigator# 32596, Sopot
  - Site Reference ID/Investigator# 32597, Sopot
  - Site Reference ID/Investigator# 43250, Wroclaw
- Romania (42):
  - Site Reference ID/Investigator# 31675, Brasov
  - Site Reference ID/Investigator# 31678, Bucharest
  - Site Reference ID/Investigator# 32568, Bucharest
  - Site Reference ID/Investigator# 32569, Bucharest
  - Site Reference ID/Investigator# 32570, Bucharest
  - Site Reference ID/Investigator# 32571, Bucharest
  - Site Reference ID/Investigator# 32098, Bucharest
  - Site Reference ID/Investigator# 32099, Bucharest
  - Site Reference ID/Investigator# 32575, Bucharest
  - Site Reference ID/Investigator# 32576, Bucharest
  - Site Reference ID/Investigator# 32577, Bucharest
  - Site Reference ID/Investigator# 32578, Bucharest
  - Site Reference ID/Investigator# 31669, Bucharest
  - Site Reference ID/Investigator# 31670, Bucharest
  - Site Reference ID/Investigator# 31671, Bucharest
  - Site Reference ID/Investigator# 31672, Bucharest
  - Site Reference ID/Investigator# 32094, Bucharest
  - Site Reference ID/Investigator# 32090, Bucharest
  - Site Reference ID/Investigator# 32091, Bucharest
  - Site Reference ID/Investigator# 32100, Cluj-Napoca
  - Site Reference ID/Investigator# 32097, Cluj-Napoca
  - Site Reference ID/Investigator# 32101, Constanța
  - Site Reference ID/Investigator# 32103, Constanța
  - Site Reference ID/Investigator# 31673, Craiova
  - Site Reference ID/Investigator# 31674, Craiova
  - Site Reference ID/Investigator# 19163, Iași
  - Site Reference ID/Investigator# 31668, Iași
  - Site Reference ID/Investigator# 32114, Iași
  - Site Reference ID/Investigator# 32115, Iași
  - Site Reference ID/Investigator# 32116, Iași
  - Site Reference ID/Investigator# 32117, Iași
  - Site Reference ID/Investigator# 32118, Iași
  - Site Reference ID/Investigator# 32119, Iași
  - Site Reference ID/Investigator# 32112, Piatra Neamţ
  - Site Reference ID/Investigator# 32572, Ploieşti
  - Site Reference ID/Investigator# 32573, Ploieşti
  - Site Reference ID/Investigator# 32574, Ploieşti
  - Site Reference ID/Investigator# 31676, Sf. Gheorghe Jud. Covasna
  - Site Reference ID/Investigator# 32104, Târgu Mureş
  - Site Reference ID/Investigator# 32105, Târgu Mureş
  - Site Reference ID/Investigator# 32108, Timișoara
  - Site Reference ID/Investigator# 32113, Timișoara
- Slovakia (3):
  - Site Reference ID/Investigator# 19164, Banská Bystrica
  - Site Reference ID/Investigator# 43262, Bratislava
  - Site Reference ID/Investigator# 43263, Košice
- Ukraine (24):
  - Site Reference ID/Investigator# 43242, Dnipro
  - Site Reference ID/Investigator# 48364, Dnipropetrovsk
  - Site Reference ID/Investigator# 31693, Donetsk
  - Site Reference ID/Investigator# 31685, Donetsk
  - Site Reference ID/Investigator# 31690, Kharkiv
  - Site Reference ID/Investigator# 31686, Kharkiv
  - Site Reference ID/Investigator# 31679, Kiev
  - Site Reference ID/Investigator# 31680, Kiev
  - Site Reference ID/Investigator# 31684, Kiev
  - Site Reference ID/Investigator# 31682, Kiev
  - Site Reference ID/Investigator# 31683, Kiev
  - Site Reference ID/Investigator# 48363, Kiev
  - Site Reference ID/Investigator# 48365, Kryvyi Rih
  - Site Reference ID/Investigator# 48366, Lviv
  - Site Reference ID/Investigator# 48367, Lviv
  - Site Reference ID/Investigator# 48368, Lviv
  - Site Reference ID/Investigator# 31689, Odesa
  - Site Reference ID/Investigator# 31694, Simferopol
  - Site Reference ID/Investigator# 43243, Uzhhorod
  - Site Reference ID/Investigator# 48369, Uzhhorod
  - Site Reference ID/Investigator# 48370, Uzhhorod
  - Site Reference ID/Investigator# 31691, Vinnitsa
  - Site Reference ID/Investigator# 31692, Zaporogzhe
  - Site Reference ID/Investigator# 48371, Zhytomyr

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigational sites in 7 countries participated in this study: Croatia, Hungary, Israel, Poland, Romania, Slovakia and Ukraine.
Pre-assignment Details: Out of 809 participants recruited, 789 were included in the statistical evaluation dataset (SES). 20 participants were not included due to no documented Humira therapy and/or missing primary diagnosis.
Groups:
- Rheumatoid Arthritis (RA): Participants with active rheumatoid arthritis
- Psoriatic Arthritis (PsA): Participants with active psoriatic arthritis
- Ankylosing Spondylitis (AS): Participants with active ankylosing spondylitis
Period: Overall Study
Arm/Group | Rheumatoid Arthritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS)
Started | 431 | 124 | 234
Completed | 324 | 95 | 166
Not Completed | 107 | 29 | 68

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS) | Total
Number analyzed (Participants) | 431 | 124 | 234 | 789
Age Continuous [Mean (Standard Deviation); unit: years] | 54.0 (11.5) | 47.8 (12.4) | 41.5 (13.0) | 49.3 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 360 | 61 | 60 | 481
  Male | 71 | 63 | 174 | 308
Disease Activity Score (DAS28) [Number; unit: participants] — DAS28 score is calculated using the number of tender and swollen joints (out of 28 counted), erythrocyte sedimentation rate (ESR) level, and the patient's global assessment of disease activity. The calculated range of DAS28 is 0.49 to 9.07, with scores below 3.2 indicating low disease activity.
  participants
    Missing | 17 | NA — This assessment was for participants with RA only, per protocol. | NA — This assessment was for participants with RA only, per protocol. | 17
    Low Disease Activity (score ≥2.6 and <3.2) | 1 | NA — This assessment was for participants with RA only, per protocol. | NA — This assessment was for participants with RA only, per protocol. | 1
    Moderate Disease Activity (score ≥3.2 and <5.1) | 37 | NA — This assessment was for participants with RA only, per protocol. | NA — This assessment was for participants with RA only, per protocol. | 37
    High Disease Activity (score ≥5.1) | 376 | NA — This assessment was for participants with RA only, per protocol. | NA — This assessment was for participants with RA only, per protocol. | 376
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score [Number; unit: participants] — BASDAI score was calculated using a questionnaire with 6 questions that participant completes by marking answers on a 10-centimeter visual analog scale with responses that range from 0 (none) to 10 (very severe) and measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 to 10.
  participants
    Missing | NA — This assessment was for participants with PsA and AS only, per protocol. | 64 | 7 | 71
    Low Disease Activity (BASDAI score <4) | NA — This assessment was for participants with PsA and AS only, per protocol. | 7 | 10 | 17
    High Disease Activity (BASDAI score ≥4) | NA — This assessment was for participants with PsA and AS only, per protocol. | 53 | 217 | 270

OUTCOME MEASURES:

1. Primary Outcome: Clinical Outcome (Disease Activity Score [DAS28] Decrease ≥1.2) After 3 Months of Humira Therapy Relative to Baseline in Participants With RA
Description: DAS28 score was calculated using the number of tender and swollen joints (out of 28 counted), erythrocyte sedimentation rate (ESR) level, and the participant's global assessment of disease activity. The calculated range of DAS28 is 0.49 to 9.07, with scores below 3.2 indicating low disease activity. A positive clinical outcome was defined as a DAS28 decrease by 1.2 or more after 3 months of Humira therapy relative to baseline.
Time Frame: Baseline, 3 months
Population: Clinical Outcome Analysis Set (COS): all participants in the SES, who had a non-missing assessment of clinical outcome at baseline and not less than one follow-up visit with a non-missing assessment of clinical outcome. In addition, patients with unclear visit schedule were excluded from the COS.
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis (RA)
Number analyzed (Participants) | 385
participants
  Missing | 56
  Positive (DAS28 Decrease ≥1.2) | 251
  Negative (DAS28 Decrease <1.2 or No Decrease) | 78

2. Primary Outcome: Clinical Outcome (Bath Ankylosing Spondylitis Disease Activity Index [BASDAI] Decrease ≥50%) After 3 Months of Humira Therapy Relative to Baseline in Participants With PsA and AS
Description: BASDAI score was calculated using a questionnaire with 6 questions that the participant completes by marking answers on a 10-centimeter visual analog scale with responses that range from 0 (none) to 10 (very severe) and measures severity of fatigue, spinal and peripheral joint pain, localized tenderness and morning stiffness. The final BASDAI score ranges from 0 to 10. A positive clinical outcome was defined as a 50% or more decrease in BASDAI score after 3 months of Humira therapy relative to baseline.
Time Frame: Baseline, 3 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS)
Number analyzed (Participants) | 52 | 216
participants
  Missing | 2 | 12
  Positive (BASDAI Decrease ≥50%) | 24 | 138
  Negative (BASDAI Decrease <50% or No Decrease) | 26 | 66

3. Secondary Outcome: Physical Function: Mean Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Baseline, and After 4, 7 and 13 Months of Humira Therapy
Description: HAQ-DI score was calculated using the standard questionnaire covering 8 category scores: Dressing and Grooming, Rising, Eating, Walking, Hygiene, Reach, Grip, and Activities. Each category score is calculated as the maximum of the scores for the questions within the category. The HAQ-DI is expressed on a scale from 0 (without any difficulty) to 3 (unable to do) representing an average score across the category. Scores for at least 6 categories are needed to compute the HAQ score. Changes to lower scores indicate improvement in physical function.
Time Frame: Baseline, 4, 7 and 13 months
Population: SES=participants fulfilling both of the following criteria: a primary diagnosis of specified rheumatic disease (RA, PsA, AS); at least one recorded Humira treatment is documented. n=number of participants with evaluable records at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Participants (RA, PsA, AS): Participants with active rheumatoid arthritis, psoriatic arthritis, or ankylosing spondylitis
Arm/Group | Rheumatoid Arthritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS) | All Participants (RA, PsA, AS)
Number analyzed (Participants) | 431 | 124 | 234 | 789
units on a scale
  Score at Baseline (n=314, 81, 106, 501) | 1.8 (0.6) | 1.5 (0.6) | 1.3 (0.6) | 1.6 (0.6)
  Score at 4 Months (n=232, 56, 76, 364) | 1.3 (0.7) | 0.8 (0.6) | 0.7 (0.5) | 1.1 (0.7)
  Score at 7 Months (n=211, 49, 63, 323) | 1.2 (0.7) | 0.7 (0.6) | 0.7 (0.6) | 1.0 (0.7)
  Score at 13 Months (n=174, 47, 31, 252) | 1.1 (0.7) | 0.8 (0.6) | 0.6 (0.5) | 1.0 (0.7)

4. Secondary Outcome: Participant Acceptability of Self-injection at Month 13 (End of Study)
Description: Participant acceptability of self-injection was assessed by the percentage of participants able to appropriately execute self-injection after initial training in the medical center, per investigator's opinion and documentation of necessity of re-training. Those participants able to self-inject also reported their experience of self-injection as convenient or inconvenient.
Time Frame: 13 months
Population: Participants in the SES with evaluable values. SES=participants fulfilling both of the following criteria: a primary diagnosis of specified rheumatic disease (RA, PsA, AS); at least one recorded Humira treatment is documented.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS) | All Participants (RA, PsA, AS)
Number analyzed (Participants) | 428 | 121 | 233 | 782
percentage of participants
  Able to Self-inject, Assessed as Convenient | 86.2 | 95.9 | 92.3 | 89.5
  Able to Self-inject, Assessed as Inconvenient | 7.2 | 0.8 | 6.4 | 6.0
  Unable to Self-inject With Need for Retraining | 0.5 | 0.0 | 0.4 | 0.4
  Unable to Self-inject Due to Disease Condition | 6.1 | 3.3 | 0.9 | 4.1

5. Secondary Outcome: Compliance With the Humira Administration Schedule at Month 13 (End of Study)
Description: Compliance with the Humira therapy was assessed by the number of missed injections among participants. Documentation of injections missed or delayed by more than 7 days was made at each study visit.
Time Frame: Month 13
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS) | All Participants (RA, PsA, AS)
Number analyzed (Participants) | 428 | 121 | 233 | 782
participants
  None | 403 | 109 | 210 | 722
  1 Injection Missed | 11 | 5 | 7 | 23
  2 Injections Missed | 0 | 3 | 8 | 11
  3 or More Injections Missed | 14 | 4 | 8 | 26

6. Secondary Outcome: Tolerability: Duration of Humira Therapy in Participants Who Discontinued Therapy
Description: Tolerability was evaluated by assessing the mean duration (in weeks) of treatment with Humira until the development of an adverse event leading to treatment discontinuation or until early discontinuation for any other reason.
Time Frame: From first treatment until study discontinuation, up to 13 months.
Population: Participants in the SES who discontinued therapy and had evaluable records. SES=participants fulfilling both of the following criteria: a primary diagnosis of specified rheumatic disease (RA, PsA, AS); at least one recorded Humira treatment is documented.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Rheumatoid Arthritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS) | All Participants (RA, PsA, AS)
Number analyzed (Participants) | 106 | 29 | 67 | 202
weeks | 28.6 (17.6) | 29.7 (19.0) | 29.9 (14.1) | 29.2 (16.7)

7. Secondary Outcome: Tolerability: Overall Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Tolerability was measured by AEs and SAEs, collected during the course of the study. See the Reported Adverse Event section for details.
Time Frame: From the time participant gave authorization to use and disclose information (or gave informed consent) until 5 half-lives following the last dose of physician-prescribed therapy. Mean (standard deviation [SD]) duration of therapy was 49.0 (16.0) weeks.
Population: SES=participants fulfilling both of the following criteria: a primary diagnosis of specified rheumatic disease (RA, PsA, AS); at least one recorded Humira treatment is documented.
Measure: Number; unit: participants
Arm/Group | Rheumatoid Arthritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS) | All Participants (RA, PsA, AS)
Number analyzed (Participants) | 431 | 124 | 234 | 789
participants
  Number of Participants with Any AE | 78 | 30 | 36 | 144
  Number of Participants with Any SAE | 18 | 4 | 5 | 27

ADVERSE EVENTS:
Time Frame: From the time participant gave authorization to use and disclose information (or gave informed consent) until 5 half-lives following the intake of the last dose of physician-prescribed treatment. Mean (SD) duration of treatment was 49.0 (16.0) weeks.
Arm/Group | Rheumatoid Arthritis (RA) | Psoriatic Arthritis (PsA) | Ankylosing Spondylitis (AS) | All Participants (RA, PsA, AS)
Serious Adverse Events (participants affected / at risk) | 18/431 | 4/124 | 5/234 | 27/789
Other Adverse Events (participants affected / at risk) | 0/431 | 0/124 | 0/234 | 0/789
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis (RA) (N=431) | Psoriatic Arthritis (PsA) (N=124) | Ankylosing Spondylitis (AS) (N=234) | All Participants (RA, PsA, AS) (N=789)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 2
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Death (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Nephrectomy (Surgical and medical procedures) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.